CLINICAL TRIAL: NCT04943783
Title: Application of Atorvastatin in the TREATment of Patients With Intracranial Unruptured Vertebrobasilar Dissecting Aneurysms
Brief Title: Atorvastatin in the TREATment of Intracranial Unruptured VertebroBasilar Dissecting Aneurysms
Acronym: ATREAT-VBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: BNI-20210601
Record Dates: First submitted 2021-05-31; First posted 2021-06-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-06

CONDITIONS: Dissecting Aneurysm of Cerebral Artery; Intramural Hematomas; Inflammation Vascular
Keywords: High resolution magnetic resonance; Atorvastatin
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin, 20mg once a day, for six months
  Interventions: Drug: Atorvastatin 20mg
- No drug (No Intervention): no drug

INTERVENTIONS:
Drug: Atorvastatin 20mg — One with the intervention (Atorvastatin, 20mg OD), 20 patients for this arm.
  Arms: Atorvastatin

SUMMARY:
This study was designed to whether there is a measurable reduction in inflammation in walls of unruptured vertebrobasilar dissecting aneurysms with atorvastatin.

DETAILED DESCRIPTION:
Unruptured vertebrobasilar dissecting aneurysms (UVBDAs) are a pathological condition of the vertebrobasilar artery caused by hypertension, atherosclerosis, and infection. Hematoma between intima and media can progressively occlude the parent artery. Thus lead to decreasing perfusion of the distal perforator vessels and even cause cerebral infarction. Even worse, ruptured VBDAs can lead to subarachnoid hemorrhage and eventually death of the patients. Thus, risk of UVBDAs rupture should be weighed, and need an individual criterion for predicting rupture in clinical decision making.

Recently, many histopathological studies indicated that inflammation may play an important role in the formation, growth, and rupture of aneurysms. High-resolution vessel wall MRI (HR-VW-MRI) has been increasingly applied in clinical practice and is the only noninvasive method for imaging the structure of the vascular wall.

Wall enhancement of an aneurysm on high resolution magnetic resonance (HRMRI) is a proven sign of inflammatory change and might predict an unsteady state of an intracranial aneurysm. Besides, a previous study has demonstrated that HR-MRI can provide valuable information, such as parameters of intramural hematomas, double lumens and intimal flaps, in the diagnosis and follow-up UVBDAs.

Statins (3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors) are widely used cholesterol-lowering drugs and are established as first-line treatments for hypercholesterolemia. In addition, statins exert pleiotropic effects to protect the vasculature. Statins can reduce the inflammation of the vessel wall and mobilize endothelial progenitor cells for aneurysmal endothelial cell repair. Statins can also inhibit the expression of several matrix metalloproteinases by smooth muscle cells and macrophages, which may be important in reducing the growth and rupture of UVBDAs.

In this study, participants with UVBDAs that are not planned for surgical treatment and has not yet ruptured, take atorvastatin daily for six months, and have a HRMRI scan before and after conservative therapy to look for the role of atorvastatin in inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 or over, male or non-pregnant female;
2. Patients have a unruptured vertebrobasilar dissecting aneurysm identified on imaging (CT, MRI or DSA)
3. Patients with wall enhancement and intramural hematomas of UVBDAs by HR-VW-MRI before treatment.
4. Patients who is able to understand the objective of the trail, agrees and signs the written informed consent form.

Exclusion Criteria:

1. The aneurysm types of non-dissecting aneurysm, such as saccular aneurysms, fusiform aneurysms and traumatic aneurysms, etc.;
2. Patients with MRI contraindications: metallic implant, contrast allergy, claustrophobia, etc.;
3. Planned treatment of the aneurysm within 6 months;
4. Several impaired liver or renal functions;
5. Retreatment of recurrent aneurysm;
6. Pregnant or lactating women;
7. Patients with malignant diseases, such as liver disease, kidney diseases, congestive heart failure, malignant tumors, etc.;
8. Poor compliance patients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
1.Change of aneurysm wall inflammation as measured by HR-VW-MRI. | 6 months
  Change of aneurysm wall enhancement index of at least 20% on HR-VM-MRI at the end of 6 months of atorvastatin 20mg daily treatment, compared to no treatment.

SECONDARY OUTCOMES:
Change of aneurysmal morphology parameter （the largest diamater） | 6 months
  Change of aneurysmal morphology parameter between pre-treatment and the 6 months follow-up periods.
Change of wall features of UVBDAs | 6 months
  Change of wall features of UVBDAs, which is intramural hematoma between pre-treatment and the 6 months follow-up periods. (The maximum diameter of the false lumen was compared)
Change of inflammatory markers in UVBDAs patients | 6 months
  Change of inflammatory markers in UVBDAs patients between pre-treatment and the 6 months follow-up periods. (CRP, TNF alpha, IL-2,6,8,10 and IL-1 beta)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Mirzat Turhon, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Data are available on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: Data are available on reasonable request.

REFERENCES:
- [Derived] Zhang Y, Wang C, Dong L, Turhon M, Kang H, Liu J, Duan Y, Tian D, Sui B, Zhang Y, Wang K, Mossa-Basha M, Yang X, Zhu C. Statins Reduce Wall Enhancement at Vessel Wall MRI in Unruptured Vertebrobasilar Dissecting Aneurysms: A Randomized Controlled Trial. Radiology. 2025 Dec;317(3):e242806. doi: 10.1148/radiol.242806. PMID 41432563
- [Derived] Turhon M, Kang H, Huang J, Li M, Liu J, Zhang Y, Wang K, Yang X, Zhang Y. Atorvastatin for unruptured intracranial vertebrobasilar dissecting aneurysm (ATREAT-VBD): protocol for a randomised, double-blind, blank-controlled trial. BMJ Open. 2022 Apr 28;12(4):e059616. doi: 10.1136/bmjopen-2021-059616. PMID 35487525